CLINICAL TRIAL: NCT03438305
Title: Role of Gastric Ultrasound in Preoperative Assessment of Gastric Volume in Longstanding Diabetic Patients. (Prospective Observational Study).
Brief Title: Role of Gastric Ultrasound in Preoperative Assessment of Gastric Volume in Diabetic Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherin Refaat, Lecturer of Anesthiology, Cairo University
Other Study IDs: N-74-2017
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group D
  Interventions: Other: sonar assessment of gastric volume in Diabetic patients
- Group N
  Interventions: Other: sonar assessment of gastric volume in Non Diabetic patients

INTERVENTIONS:
Other: sonar assessment of gastric volume in Diabetic patients — assessment of gastric volume in Diabetic Patients
  Groups: Group D
Other: sonar assessment of gastric volume in Non Diabetic patients — assessment of gastric volume in Non- Diabetic Patients
  Groups: Group N

SUMMARY:
Background :An important risk factor for aspiration is gastric volume, determined in large part by gastric emptying. Unfortunately, measuring gastric volume over time is not easy, and scintigraphy has remained the gold standard technique for many years. Ultrasound has progressively emerged as a useful substitute due to its reduced cost and ease of performance Objectives:Assess whether ultrasonographic measurement of antral cross sectional area (CSA) can be used reliably for the diagnosis of risk stomach which defined by a gastric content volume at risk of clinical consequences for pulmonary aspiration (i.e., presence of solid particles and/or gastric fluid volume >1.5 ml/kg) during the preoperative period in longstanding diabetic patients.

Study population :

* -Longstanding diabetic patients (group D)
* -Non diabetic patients (group N) Study Design : Prospective observational study This study will be conducted at Kasr alainy Hospital; Faculty of Medicine, Cairo University.Patients scheduled for elective operations need General Anesthesia (GA) with endotracheal intubation in theatre of general surgery Preoperative ultrasound to assess gastric residual volume then general anesthesia induction will be Modified Rapid-sequence Induction as follow; Group (D)/(N) : propofol 2-3mg/kg and fentanyl 1 µg/Kg followed by Rocuronium 0.6-1.2 mg/kg.

Suction of Gastric Contents by Nasogastric tube (18 french) will be inserted First set of analysis will be comparing preoperative US findings in 2 groups.

Second set of analysis will be finding correlation between US findings and suction volume in two groups.

Outcome parameters: To assess the residual gastric volume in longstanding diabetic patients compared to non diabetic patients.

Sample Size ; was calculated as 48 patients (24) in each group.

ELIGIBILITY:
Inclusion Criteria:

* Ages from 40 to 60 years old.
* American Society of Anesthiologist (ASA) II.
* Diabetic patients with longstanding duration(more than 6 years).

Exclusion Criteria:

* Age <40,>60 years .
* Pregnant female
* Obese patients (BMI ≤40)
* Patients with Gastric Intestinal Tract (GIT) diseases affect gastric emptying.
* Diabetic patients less than 6 years.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Diabetic patients with long standing diabetis ( more than 6 years) so , it may affect gastric nerve supply.
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
assessment of residual gastric volume in longstanding diabetic patients | intra-operative
  To assess the residual gastric volume in longstanding diabetic patients compared to non diabetic patients

SECONDARY OUTCOMES:
correlation between preoperative gastric US findings and fasting hours in both groups | intraoperative
  To correlate between preoperative gastric US findings and fasting hours in both groups to confirm delayed gastric emptying in diabetic group.

REFERENCES:
- [Derived] Sabry R, Hasanin A, Refaat S, Abdel Raouf S, Abdallah AS, Helmy N. Evaluation of gastric residual volume in fasting diabetic patients using gastric ultrasound. Acta Anaesthesiol Scand. 2019 May;63(5):615-619. doi: 10.1111/aas.13315. Epub 2019 Jan 4. PMID 30609007